CLINICAL TRIAL: NCT00217776
Title: School-based Approaches to Help Pre-teens Manage Asthma
Acronym: DMSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Noreen M. Clark, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 288; R01HL068654-04 (NIH)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Open Airways Educational Intervention (Active Comparator): Children in this arm will receive the Open Airways educational program which is an evidenced based asthma educational program for children, developed by the investigator.
  Interventions: Behavioral: Open Airways Educational Intervention
- Open Airways and Peer Asthma Action Intervention Education (Active Comparator): Children in this arm will receive BOTH the Open Airways asthma education program and the Peer Asthma Action education program.
  Interventions: Behavioral: Open Airways Educational Intervention; Behavioral: Peer Asthma Action Educational Intervention
- Control Arm (No Intervention): Children in the Control Arm will be interviewed in person at baseline, 12 month and 24 months.

INTERVENTIONS:
Behavioral: Open Airways Educational Intervention
  Other Names: A 6 week asthma educational self management program for middle school students.
  Arms: Open Airways Educational Intervention; Open Airways and Peer Asthma Action Intervention Education
Behavioral: Peer Asthma Action Educational Intervention
  Other Names: Peer Asthma Action Educational Intervention is a peer led training program for children in multiple grades teaching them about asthma and asthma management.
  Arms: Open Airways and Peer Asthma Action Intervention Education

SUMMARY:
This random trial will deploy 2 interventions and a control group with eleven and twelve year old, low income, African American students in middle schools in Detroit, MI. The goals are to determine if 1) a self-management program focused on pre-teen capabilities designed for middle schools produces desired outcomes, and 2) if the program, enhanced by a peer component, improves upon outcomes. Outcomes of interest are symptom experience, quality of life, self-management, and school grades.

DETAILED DESCRIPTION:
BACKGROUND:

To date, no data provide information on the effects of middle school based interventions for pre-teens with asthma or the advantages of an approach that recognizes the importance of peer influence on pre-teen's asthma behavior. Interventions to reach low income minority populations are particularly needed.

DESIGN NARRATIVE:

If only one primary outcome is to be specified, it would be asthma morbidity, as evident in asthma symptoms. Data to assess outcomes will be collected at baseline, and 12 and 24 months post program through parent interviews and student surveys.

Additional primary outcomes listed in the protocol include: Asthma related quality of life, disease management behavior and academic performance.

Secondary outcomes include: peer support, school attendance, physical activity, health care use, and smoking behavior.

ELIGIBILITY:
Children identified for this research will be a sample of 6th grade students enrolled in 19 public middle schools in Detroit, Michigan who meet the following criteria: 1) attend a participating school, 2) be 11-12 years old at the time of entry into the study (enrolled in 6th grade) and 3) based on NAEPP guidelines (a) have a diagnosis of asthma and have active asthma symptoms and/or have received a prescription for asthma medications in the last year, or (b) report the presence of 3 of 5 non-exercise related asthma symptoms in the last year on five or more occasions, or (c) report two or more exercise related asthma symptoms in the past year on five or more occasions, or (d) have a severity classification of persistent disease (mild, moderate, severe) based on night time questions, and 4) have returned a signed parental consent form.

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1292 (Actual)
Dates: Start 2003-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Health Care Use Data | At Baseline, 12 month and 24 months
  health care use will be self reported in the telephone interviews with parents at baseline, 12 months and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Noreen M. Clark, PhD, Principal Investigator — University of Michigan School of Public Health